CLINICAL TRIAL: NCT06503562
Title: The Effect of Central Nervous System Focused Treatment Program in Chronic Nonspecific Neck Pain -Randomised Controlled Trial
Brief Title: Chronic Nonspecific Neck Pain and Central Nervous System Focused Treatment Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assoc, Prof. Nuray Alaca, Head of department Physiotherapy and Rehabilitation, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATADEK-2024-9/341
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Neck Pain; Chronic Pain Syndrome; Rehabilitation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Physiotherapy Program (Other)
  Interventions: Other: Classical Physiotherapy
- Traditional Physiotherapy Program and central nervous system focused treatment program (Experimental)
  Interventions: Other: central nervous system focused treatment program; Other: Classical Physiotherapy

INTERVENTIONS:
Other: central nervous system focused treatment program — Pain neuroscience education, breathing exercises and relaxation exercises with guided imagery
  Arms: Traditional Physiotherapy Program and central nervous system focused treatment program
Other: Classical Physiotherapy — All participants will receive conventional physiotherapy five days a week for one month. Transcutaneous electrical nerve stimulation, 15 min hotpack will be applied to the neck and back. Afterwards, mobilisations to the cervical and thoracic spine joints and myofascial release to the upper trapezius muscle will be applied. The patient will be given 3X10 neck active range of motion exercises to do at home every day and self stretches to the muscles in the neck region (SCM, upper trapezius, scalene and pectoral) according to the patient's condition. After the first week, strengthening exercises with isometric and resistive isotonic exercises will be given to the neck and upper back muscles gradually increasing. Patients will not be given any medication and will be asked not to use any medication.

SUMMARY:
Neck pain is one of the most common musculoskeletal pain disorders secondary to low back pain. Pharmacological and non-medical treatments such as physiotherapy are applied in its treatment. Patients with chronic nonspecific neck pain (CNSP) can be treated with various interventions such as drug therapy, manual therapy, heat and exercise. However, it is also reported that chronic pain occurs as a result of neuroplasticity, that is, the brain learning pain through the central synthesis mechanism in the central nervous system. For this reason, although the importance of central nervous system-oriented therapies is increasing day by day, this system-oriented therapies are still ignored in clinics. Therefore, in this master's thesis study, it is aimed to investigate the effects of central nervous system-focused therapies (pain neuroscience education, breathing exercises and relaxation exercises with guided imagery) on pain, range of motion, functional status, pain-related fear, anxiety, depression and quality of life in addition to traditional physiotherapy applied to patients with CNSP.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with nonspecific neck pain by a doctor,
* To be between the ages of 18-65,
* Having neck pain for more than 3 months
* No previous neck or shoulder surgery,
* No shoulder pain due to any cause,
* A tumour or inflammatory disease underlying the neck pain not to be found,
* A clinically underlying stenosis or discogenic problem not to be present.
* Negative results from the following clinical examination tests;

  * Spurling test,
  * Lhermitte test,
  * Cervical distraction test,
  * Adson test,

Exclusion Criteria:

* Not meeting the inclusion criteria,
* Positive neurological examination (positive motor presence, reflex or sensory abnormalities indicating spinal root compression) or abnormal neurological findings related to nerve compression in the upper limb
* Systemic rheumatological or metabolic diseases or cancer
* Refusal to participate in the study,
* Failure to complete treatment,
* Having any neurological problem
* Severe psychological illnesses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-11-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
The Numerical Rating Scale (NPRS-11) | Change from baseline range of motion at 4th week
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
Range of Motion | Change from baseline range of motion at 4th week
  CROM device will be used. The active range of motion of each individual will be measured and measured in accordance with the manufacturer's procedures
Pressure Pain Threshold | Change from baseline range of motion at 4th week
  A digital pressure algometer will be applied to the web space of the foot opposite the trigger point. Participants are instructed to say "stop" or "pain" so the stimulus can be terminated "when the sensation first transitions from pressure to pain" (pain threshold).
Neck disability index | Change from baseline range of motion at 4th week
  Since some parts of the 10-item questionnaire could not be answered by the patients (driving, working life), the average neck disability index score will be calculated by dividing the total score by the number of questions answered. The scoring is between 0 and 50. 0 points means the best result, 50 points means the worst result. 0 - 4 points; no disability, 5 - 14 points; mild disability, 15 - 24 points; moderate disability, 25 - 34 points; severe disability, > 35 points; complete disability
Pain Catastrophizing Scale | Change from baseline range of motion at 4th week
  Catastrophobia one of the cognitive and emotional outcomes of chronic pain, is an important concept related to the perception of pain. Catastrophobic people tend to feel pain more severe than it actually is. The Pain Catastrophobia Scale consists of 13 items and assesses the frequency of concerns about the perception and persistence of existing pain. It has 3 subheadings: helplessness, magnification and rumination. It is scored as never (0) and always (4). The person can score a total of 52 points
Fear avoidance belief questionnaire | Change from baseline range of motion at 4th week
  Fear avoidance belief questionnaire is a questionnaire based on the fear-avoidance model of exaggerated pain perception. The FABQ measures patient's fear of pain and consequent avoidance of physical activity (PA) because of their fear.There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs. There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24)

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Change from baseline range of motion at 4th week
  It containing 19 self-rated questions searching the sleep quality during the previous month. It has seven components as subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction.
  Each component is scored from 0 to 3, and the Global Pittsburgh Quality of Sleep (PQS) score is the sum of the scores of the seven components that is between 0 and 21. The higher Global PQS scores indicate poor sleep quality and the cut off score for poor sleep is 5 and over.
SF 12 Quality of life | Change from baseline range of motion at 4th week
  A health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health.Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. A score of 50 or less on the physical-quality of life 12 has been recommended as a cut-off to determine a physical condition; while a score of 42 or less on the mental quality of life may be indicative of 'clinical depression.
Hospital Anxiety and Depression Scale | Change from baseline range of motion at 4th week
  Hospital Anxiety and Depression Scale questionnaire. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
Central Sensitization Scale | Change from baseline range of motion at 4th week
  Central Sensitization Scale, which can be applied in the presence of chronic pain, is used in central sensitization syndromes. It consists of two parts. Part A of the scale includes a Likert scale (0-4 points) that questions health-related symptoms. This section is scored from 0 to 100, with higher numbers being associated with a higher degree of central sensitization. Scores of 40 and above indicate the presence of central sensitization. In section B, it questions whether any of the central sensitization syndromes have been diagnosed before.
Global Rating of Change scale (Patient Satisfaction) | Change from baseline range of motion at 4th week
  Patient satisfaction regarding improvement in shoulder function will be evaluated by the Global Rating of Change scale. All participants will be asked to rate their condition after a six-week intervention period compared to baseline by indicating whether they have improved significantly, improved slightly, unchanged, deteriorated slightly, or deteriorated significantly between -3 to +3, with a higher value indicating better condition in this study.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acibadem University, Istanbul
  - Nuray ALACA, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided